CLINICAL TRIAL: NCT00336206
Title: Subcutaneous Injection, Low Dose Alemtuzumab for Consolidation and Maintenance of Patients in Clinical Response After Having Achieved Partial or Complete Remission After 1st or 2nd Line Anti-Tumor Therapy for B-Cell CLL
Brief Title: Low Dose Alemtuzumab for Consolidation and Maintenance of Patients With B-Cell Chronic Lymphocytic Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tawam Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 39338
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2006-07-25 (Estimated); Status verified 2006-06

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
Keywords: Low dose Alemtuzumab; Chronic lymphocytic leukemia; B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab

SUMMARY:
The aim of the study is to evaluate if the treatment with Alemtuzumab (after I or II line chemotherapy) administered for 6 weeks followed by 4 months maintenance treatment compared to a control group can reduce disease activity/residual disease and thereby delay the reoccurrence of the CLL disease.

DETAILED DESCRIPTION:
Fludarabine (F) alone or in combination with cyclophosphamide (FC) is not a curative treatment for patients with CLL, all patients will eventually relapse. Therefore there is a medical need to look for consolidation followed by maintenance therapies which are able to prolong response duration or which can shift anti-tumor therapy induced partial remissions to complete remissions or eradicate minimal residual disease in complete - but still PCR-positive - responders.

There is no standard consolidation therapy available at the moment and the role of consolidation in CLL has recently been acknowledged as a research field of major importance in B-CLL (Schering global advisory board meeting, Lisbon Nov 2005). Possible treatment options are high-dose chemotherapy followed by autologous stem cell transplantation (the role of which however remains uncertain with lack of worldwide consensus) or monoclonal antibody therapy against antigens expressed by CLL cells. Alemtuzumab is directed against the CD52-antigen which is present in high density on CLL cells and may therefore be most suitable for treatment of residual disease.

Alemtuzumab has shown significant remission rates in patients with fludarabine refractory CLL and sub analysis revealed a very high effectiveness of the antibody in clearing CLL cells from peripheral blood and bone marrow. These findings suggest that Alemtuzumab might be an ideal candidate to eliminate minimal residual disease in a post-remission treatment after anti-tumor therapy and to be used as maintenance therapy. The efficacy of Alemtuzumab as consolidation therapy in CLL can easily be measured. There is evidence from several studies that treatment with Alemtuzumab does not have a negative impact on stem cell mobilization. Therefore, autologous stem cell transplantation still remains as a further treatment option for those patients who still have detectable disease after primary cytoreduction followed by consolidation therapy with Alemtuzumab.

Side effects of s.c. Alemtuzumab in heavily pretreated patients with advanced disease are tolerable and manageable. Data have suggested that the safety profile of this antibody is even more favorable in less pretreated patients and the GCLLSG study suggests that a wash-out period of more than 8 weeks and possibly also a lower dose is necessary to avoid severe infectious problems. Campath administration started after a 2-month wash out period after Fludarabine was shown to be feasible and good tolerated. Based on the collective data obtained from other pilot or phase II studies, a subcutaneous consolidation dose of 30 mg once weekly in previously treated and untreated CLL patients after an induction with Fludarabine combination seems to be a safe and effective dose.

The proposed study aims to evaluate the efficacy of low dose treatment with Alemtuzumab with regard to the following questions: Does consolidation therapy with low dose Alemtuzumab result in a prolonged time to disease progression in comparison to patients who do not receive further treatment? Is it possible to turn a PR into a CR? Does maintenance therapy with Alemtuzumab translate into a progression-free survival benefit compared to patients with no further treatment? How is the safety profile in patients treated with low dose Alemtuzumab as MRD elimination and as maintenance therapy?

ELIGIBILITY:
Inclusion Criteria:

* B-CLL diagnosis taken consideration of NCI criteria.
* In case of CR: positive MRD status
* At least achieving a PR to the last line of antitumor therapy given and than at least PR is still present after a follow-up of 3-6 months after the last antitumor course (wash-out period)
* Age >18 years and < 75 years.
* WHO performance status 0-II.
* ANC ≥1.0 x 109/L
* Platelet count ≥50 x 109/L
* Negative pregnancy test in fertile females
* Anticipated life expectancy ≥ 12 months
* Signed informed consent
* Fertile men or women of childbearing potential using adequate contraception (oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile)

Exclusion Criteria:

* Elapsed time of less than 3 months or more than 6 months since last dose of previous antitumor therapy
* Previous Alemtuzumab administration.
* Contraindication for Alemtuzumab
* More than 2 previous treatment regimens
* SD or PD on last antitumor therapy
* Persistent CLL symptoms in clinical need of further antitumor therapy
* History of severe pneumocytis carinii infection (PCP)
* HIV positive
* Active hepatitis or a history of prior viral hepatitis B or hepatitis C, or positive hepatitis B serologies without prior immunization
* Active viral, fungal or bacterial infection.
* Active autoimmune hemolytic anemia or active autoimmune thrombocytopenia.
* Severe concurrent diseases or mental disorders.
* Significant renal dysfunction ( serum creatinine ≥150 µmol/l or creatinine clearance < 30 ml/min)
* Significant hepatic dysfunction (total bilirubin or transaminases >2 times ULN)
* Pregnancy or lactation.
* Active secondary malignancy.
* Participating in other clinical trials.
* Transformation to aggressive B-cell malignancy (e.g., large B-cell lymphoma, Richter's syndrome, or prolymphocytic leukemia (PLL);
* Bulky disease requiring anti-tumor therapy.
* Planned or previous BMT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-07; Study Completion 2009-10

PRIMARY OUTCOMES:
To determine the Time to Treatment Failure (TTF)

SECONDARY OUTCOMES:
To evaluate Complete Remission (CR) rate.
To evaluate Partial Response (PR) rate.
Minimal Residual Disease (MRD) evaluated with flow-cytometry ("MRD flow panel") in patients with CR
To determine Overall Response Rate (ORR).
To evaluate duration of response.
To evaluate safety

CONTACTS AND LOCATIONS:
Overall Officials: Jorgen Kristensen, MD PhD, Principal Investigator — Department of Oncology